CLINICAL TRIAL: NCT00719862
Title: Randomized, Double Blind, Placebo-Controlled Trial of the Safety and Efficacy of MP03-036 in Patients With Seasonal Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety & Effectiveness of a Nasal Spray to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Harry Sacks, MD Vice President, Medical and Scientific Affairs
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP439
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2010-01-28 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Nasal Spray (Placebo Comparator): 0mg Placebo Nasal Spray
  Interventions: Drug: Placebo nasal spray
- 0.15% azelastine hydrochloride nasal spray (Active Comparator): 0.15% azelastine hydrochloride
  Interventions: Drug: 0.15% azelastine hydrochloride Nasal Spray

INTERVENTIONS:
Drug: Placebo nasal spray — Placebo
  Arms: Placebo Nasal Spray
Drug: 0.15% azelastine hydrochloride Nasal Spray — 0.15% azelastine hydrochloride 822 mcg
  Other Names: astepro 0.15%
  Arms: 0.15% azelastine hydrochloride nasal spray

SUMMARY:
The Purpose of this study is to determine if one allergy medication (0.15% azelastine hydrochloride) is more effective than Placebo alone

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 12 years of age and older with a 2 year history of moderate to severe seasonal allergic rhinitis
* Must be in generally good health
* Must meet minimum symptom requirements, as specified in the protocol
* Must be willing and able to provide informed consent and to participate in all study procedures
* Positive skin test to a prevalent fall allergen

Exclusion Criteria:

* On focused Nasal Examination, the presence of any nasal mucosal erosion, nasal ulceration, or nasal septal perforation at either the screening visit or randomization visit will disqualify the subject from the study.
* Other nasal disease(s)likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa, clinically significant polyposis, or nasal structural abnormalities.
* Nasal Surgery or sinus surgery within the previous year
* Chronic sinusitis-more than 3 episodes a year
* Planned travel outside of the study area during the study period
* The use of any investigational drug within 30 days prior to screening. No investigational products are permitted for use during the conduct of the study.
* Presence of any hypersensitivity to drugs similar to azelastine and to either sorbital or sucralose (Splenda brand sweetener)
* Women who are pregnant or nursing
* Women of childbearing potential who are not abstinent or not practicing medically acceptable method of contraception
* Respiratory tract infection within 14 days prior to screening
* Respiratory tract infections requiring antibiotic treatment 14 days prior to screening
* Asthma (with the exception of mild, intermittent asthma). Subjects with mild, intermittent asthma who only require short-acting inhaled bronchodilators (not for more often tha twice a week) and who do not have nocturnal awakening as a result of asthma are eligible for enrollment
* Significant pulmonary disease including COPD
* Clinically significant arrythmia or symptomatic cardiac conditions
* A known history of alcohol or drug abuse within the last 2 years
* Existence of any surgical or medical condition or physical laboratory findings, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug; that might significantly affect the subject's ability to complete this trial; or their safety in this trial
* Clinically relevant abnormal physical findings which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (34):
- United States (34):
  - Allergy and Asthma Specialist Medical Group, Huntington Beach, California
  - Allergy, Asthma and Respiratory Care medical Center, Long Beach, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Cntr, San Jose, California
  - Bensch Research Associates, Stockton, California
  - Colorado Allergy and Asthma centers, PC, Lakewood, Colorado
  - University of South Florida, Tampa, Florida
  - Aeroallergy Research Laboratories of Savannah, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Atlanta Allergy and Asthma Clinic, Woodstock, Georgia
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Kansas City Allergy and Asthma, Overland Park, Kansas
  - RX R+D, Metairie, Louisiana
  - Chesapeake Clinical Research, Inc, Baltimore, Maryland
  - Institute for Asthma and Allergy PC, Wheaton, Maryland
  - Clinical Research Institute, Plymouth, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - Midwest Allergy and Asthma Clinic, Omaha, Nebraska
  - The Asthma and Allergy Center, Papillion, Nebraska
  - Las Vegas Physicians Research Group, Henderson, Nevada
  - Allergy and Asthma Research NJ inc, Mount Laurel, New Jersey
  - Allergy Consultants PA, Verona, New Jersey
  - AAIR Research Center, Rochester, New York
  - OIAA Clinical Research, LLC, Edmond, Oklahoma
  - Asthma and Allergy Research Associates, Chester, Pennsylvania
  - Valley Clinical Research, Easton, Pennsylvania
  - UPMC-ENT, Pittsburgh, Pennsylvania
  - Asthma, Nasal Disease & Allergy Research Center of New England, Providence, Rhode Island
  - Pharmaceutical Research & Consulting Inc, Dallas, Texas
  - Jane Lee, MD, PA Research Center, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - Advanced Healthcare, SC, Milwaukee, Wisconsin
  - Allergy and Asthma Center of Michigan, Novi, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First observation: August 20, 2007 Last observation: November 14, 2007
Pre-assignment Details: Subjects participated in a 7 day screening period to Identify appropriate subjects based on symptom scores.
Groups:
- Placebo: Placebo Nasal Spray/2 sprays per nostril once daily for 14 days
- Astepro 0.15%: 0.15% azelastine hydrochloride Nasal Spray/2sprays per nostril once daily for 14 days
Period: Overall Study
Arm/Group | Placebo | Astepro 0.15%
Started | 242 | 239 (1 subject was randomized in error)
Completed | 234 | 233
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 3 | 0
Not completed — Non-Compliance | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Astepro 0.15% | Total
Number analyzed (Participants) | 242 | 238 | 480
Age, Categorical [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    <=18 years | 29 | 22 | 51
    Between 18 and 65 years | 205 | 213 | 418
    >=65 years | 8 | 3 | 11
Age Continuous [Mean (Standard Deviation); unit: years] — Number of participants based on ITT population
  years | 35.3 (13.91) | 35.5 (13.53) | 35.4 (13.71)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants is based on ITT population
  Participants
    Female | 162 | 154 | 316
    Male | 80 | 84 | 164
Region of Enrollment [Number; unit: participants] — Participants are based on ITT population
  participants
    United States | 242 | 238 | 480

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12-hour Reflective Total Nasal Symptom Score (AM and PM Combined)at 14 Days
Description: reflective total nasal symptom score consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline and 14 days
Measure: Least Squares Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 242 | 238
scores on a scale
  Baseline symptom score | 17.72 (3.310) | 17.74 (3.540)
  Overall change from baseline | -2.55 (4.195) | -3.60 (4.469)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p = 0.005, ANOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.05, 95% CI [-1.80 to -0.31], Standard Deviation 0.3782

2. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Nasal Symptom Score (tNSS) (AM) for the Entire 14-day Study Period Compared to Placebo
Description: End of 24 hour dosing interval: This endpoint is change from baseline in instantaneous tNSS for the 14-day study period compared to placebo to observe if the duration of efficacy lasts 24 hours on a day to day basis. Instantaneous tNSS consists of runny nose, itchy nose, nasal congestion, and sneezing. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and baseline as a covariate.
Time Frame: baseline and 14 days
Measure: Least Squares Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 242 | 238
scores on a scale | -1.05 (2.059) | -1.35 (2.320)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p = 0.112, ANOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Median Difference (Final Values) = -0.2987, 95% CI [-0.67 to 0.07], Standard Deviation 0.1881

3. Secondary Outcome: Change From Baseline in 12 Hour Instantaneous Total Nasal Sytmptom Score (AM and PM Combined)at 14 Days
Description: instantaneous (subjects rate how they feel "right now") total nasal symptom score consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline and 14-days
Measure: Least Squares Mean (Standard Deviation); unit: total nasal symptom score
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 242 | 238
total nasal symptom score
  Baseline symptom score | 16.39 (3.936) | 16.23 (4.528)
  Overall change from baseline | -2.16 (4.141) | -3.03 (4.518)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Test type: Superiority or Other; p = 0.023, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.8617, 95% CI [-1.61 to -0.12], Standard Deviation .3803

4. Secondary Outcome: Change From Baseline in 12-hour Reflective SSCS for the Entire 14-day Study Period Compared to Placebo (Am and PM Combined)
Description: Reflective secondary symptom scores (SSCS) (post-nasal drip, itchy eyes, cough and headacdhe) were assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible SSCS score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline and 14-days
Measure: Least Squares Mean (Standard Deviation); unit: Refecltive secondary symptom score
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 242 | 238
Refecltive secondary symptom score
  Baseline SSCS | 13.55 (5.024) | 13.03 (5.408)
  Change in baseline to Day 14 | -1.72 (3.728) | -2.46 (3.877)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Change in baseline; Test type: Superiority or Other; p = 0.025, ANOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -0.7395, 95% CI [-1.39 to -0.09], Standard Deviation 0.3305

5. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)at 14 Days
Description: A 28-item RQLQ was completed on Day 1 and Day 14 or Early temination. The RQLQ consists of 7 domains rated on a 7 point scale with 0 being not troubled by the allergy symptoms, and 6 being extremely troubled/all of the time.
  Total overall score is not calculated by adding all subscales scores for an overall score. Domain score will be calculated from the mean score of all items in the domain. Overall score will be calculated from the mean score of all items.
Time Frame: baseline and 14 Days
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 242 | 238
Units on a scale
  Baseline: Overall | 3.51 (0.996) | 3.42 (1.101)
  Change from Baseline:Overall | -0.71 (1.172) | -0.92 (1.058)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.15%; Change from baseline; Test type: Superiority or Other; p = 0.051, ANOVA

6. Secondary Outcome: Change From Baseline on Direct Visual Nasal Exams at 14 Days
Description: Examination of head and neck (scale: None, Mild, Moderate, Severe) for Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal erythema, Mucosal Bleeding, and Crusting of mucosa. Nasal irratation was rated: 0 = None,Grade 1A = focal irritation, Grade 1B = superficial mucosal erosion, Grade 2 = moderate mucosal erosion, Grade 3 = ulceration, Grade 4 = septal perforation
Time Frame: baseline and 14 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Astepro 0.15%
Number analyzed (Participants) | 242 | 238
Participants
  Epistaxis: screening - None (n = 242, 239) | 239 | 234
  Epistaxis: screening - Mild (n = 242, 239) | 3 | 5
  Epistaxis: screening - Moderate (n = 242, 239) | 0 | 0
  Epistaxis: screening - Severe (n = 242, 239) | 0 | 0
  Epistaxis: Day 14/ET - None (n = 241, 237) | 235 | 233
  Epistaxis: Day 14/ET - Mild (n = 241, 237) | 6 | 4
  Epistaxis: Day 14/ET - Moderate (n = 241, 237) | 0 | 0
  Epistaxis: Day 14/ET - Severe (n = 241, 237) | 0 | 0
  Irritation: screening - None (n = 242, 239) | 230 | 223
  Irritation: screening - Grade 1A (n = 242, 239) | 11 | 16
  Irritation: screening - Grade 1B (n = 242, 239) | 1 | 0
  Irritation: screening - Grade 2 (n = 242, 239) | 0 | 0
  Irritation: screening - Grade 3 (n = 242, 239) | 0 | 0
  Irritation: screening - Grade 4 (n = 242, 239) | 0 | 0
  Irritation: Day 14/ET - None (n = 241, 237) | 227 | 218
  Irritation: Day 14/ET - Grade 1A (n = 241, 237) | 13 | 17
  Irritation: Day 14/ET - Grade 1B (n = 241, 237) | 1 | 2
  Irritation: Day 14/ET - Grade 2 (n = 241, 237) | 0 | 0
  Irritation: Day 14/ET - Grade 3 (n = 241, 237) | 0 | 0
  Irritation: Day 14/ET - Grade 4 (n = 241, 237) | 0 | 0
  Mucosal Edema: screening - None (n =242, 239) | 27 | 27
  Mucosal Edema: screening - Mild (n =242, 239) | 65 | 67
  Mucosal Edema: screening - Moderate (n =242, 239) | 109 | 104
  Mucosal Edema: screening - Severe (n =242, 239) | 41 | 41
  Mucosal Edema: Day 14/ET - None (n = 241, 236) | 40 | 31
  Mucosal Edema: Day 14/ET - Mild (n = 241, 236) | 102 | 102
  Mucosal Edema: Day 14/ET - Moderate (n = 241, 236) | 76 | 77
  Mucosal Edema: Day 14/ET - Severe (n = 241, 236) | 23 | 26
  Nasal Discharge: screening - None (n= 242, 239) | 26 | 50
  Nasal Discharge: screening - Mild (n= 242, 239) | 120 | 106
  Nasal Discharge: screening - Moderate (n= 242, 239 | 76 | 71
  Nasal Discharge: screening - Severe (n= 242, 239) | 10 | 12
  Nasal Discharge: Day 14/ET - None (n= 241, 237) | 81 | 70
  Nasal Discharge: Day 14/ET - Mild (n= 241, 237) | 119 | 121
  Nasal Discharge: Day 14/ET - Moderate (n= 241, 23 | 40 | 39
  Nasal Discharge: Day 14/ET - Severe (n= 241, 237) | 1 | 7
  Mucosal Erythema: screening - None (n= 242, 239) | 124 | 113
  Mucosal Erythema: screening - Mild (n= 242, 239) | 74 | 73
  Mucosal Erythema: screening - Moderate (n= 242, | 39 | 51
  Mucosal Erythema: screening - Severe (n= 242, 239 | 5 | 2
  Mucosal Erythema: Day 14/ET - None (n= 241, 237) | 146 | 142
  Mucosal Erythema: Day 14/ET - Mild (n= 241, 237) | 64 | 58
  Mucosal Erythema: Day 14/ET - Moderate (n= 241, 23 | 28 | 33
  Mucosal Erythema: Day 14/ET - Severe (n= 241, 237) | 3 | 4
  Mucosal Bleeding: screening - None (n= 242, 239) | 237 | 233
  Mucosal Bleeding: screening - Mild (n= 242, 239) | 4 | 6
  Mucosal Bleeding: screening - Moderate (n= 242, 23 | 1 | 0
  Mucosal Bleeding: screening - Severe (n= 242, 239) | 0 | 0
  Mucosal Bleeding: Day 14/ET - None (n= 241, 237) | 234 | 233
  Mucosal Bleeding: Day 14/ET - Mild (n= 241, 237) | 7 | 4
  Mucosal Bleeding: Day 14/ET - Moderate (n= 241, 23 | 0 | 0
  Mucosal Bleeding: Day 14/ET - Severe (n= 241, 237) | 0 | 0
  Crusting of Mucosa: screening - None (n= 242, 239) | 218 | 214
  Crusting of Mucosa: screening - Mild (n= 242, 239) | 22 | 23
  Crusting of Mucosa:screening Moderate (n= 242,239) | 2 | 2
  Crusting of Mucosa: screening Severe (n= 242, 239) | 0 | 0
  Crusting of Mucosa: Day 14/ET - None (n= 241, 237) | 231 | 221
  Crusting of Mucosa: Day 14/ET - Mild (n= 241, 237) | 8 | 12
  Crusting of Mucosa: Day14/ETModerate (n= 241,237) | 2 | 4
  Crusting of Mucosa: Day 14/ET Severe (n= 241, 237) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Astepro 0.15%
Serious Adverse Events (participants affected / at risk) | 0/242 | 0/238
Other Adverse Events (participants affected / at risk) | 11/242 | 17/238
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=242) | Astepro 0.15% (N=238)
Dysgusia (Nervous system disorders) | 2 (2) | 8 (8)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, joint publication is required to assure that the initial publication is based on all data from all sites and investigators participating in these studies agree not to present data gathered individually or by subgroup centers before the initial publication unless jointly agreed by all other investigators and the sponsor. authorship will be determined by mutual agreement.